CLINICAL TRIAL: NCT02364076
Title: Pembrolizumab (MK-3475) and Epacadostat (INCB024360) in Thymic Carcinomas
Brief Title: Pembrolizumab and Epacadostat in Patients With Thymic Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Georgetown University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-1315
Record Dates: First submitted 2015-02-10; First posted 2015-02-16 (Estimated); Results first posted 2019-12-13 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2018-11

CONDITIONS: Thymic Carcinoma; Thymus Neoplasms; Thymus Cancer
Keywords: Pembrolizumab; Epacadostat
MeSH Terms: conditions — Thymoma; Thymus Neoplasms | interventions — pembrolizumab; epacadostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab and Epacadostat (Experimental): Pembrolizumab 200 mg intravenously every 3 weeks Epacadostat 100mg by mouth taken daily
  Interventions: Drug: Pembrolizumab; Drug: Epacadostat

INTERVENTIONS:
Drug: Pembrolizumab — Administration of 200 mg MK-3475 once every 3 weeks
  Other Names: Keytruda; MK-3475
Drug: Epacadostat — 100mg taken by mouth twice daily
  Other Names: INCB024360

SUMMARY:
This is a non-randomized clinical trial in patients with thymic carcinomas who failed prior systemic therapy. All subjects will receive pembrolizumab and epacadostat treatment in three week cycles until unacceptable toxicity, death, progressive disease or withdrawal.

DETAILED DESCRIPTION:
The amended phase II study of pembrolizumab and epacadostat is for thymic carcinoma patients who recurred after at least one prior chemotherapy regimen. The primary endpoint is response rate; secondary endpoints are Progression-Free Survival, Overall Survival and treatment tolerability. Responses will be assessed according to RECIST 1.1; progression-free survival is defined as time between start of treatment and tumor progression or death; survival is the time between start of treatment and death. Furthermore exploratory studies will be performed on archival tumor material (PDL-1 expression, next-generation sequencing), and fresh biopsies (culturing; next-generation sequencing).

ELIGIBILITY:
Inclusion Criteria:

1. Histologic confirmation of thymic carcinoma (WHO Classification, See Appendix 12.1)
2. Advanced disease (Masaoka staging, See Appendix 12.2) not amenable to curative treatment.
3. At least 1 prior line of chemotherapy.
4. Progression of disease must be documented prior to study entry.
5. Absence of any autoimmune syndrome typically associated with thymomas but not thymic carcinomas (myasthenia gravis, pure red cell aplasia, etc.).
6. Be willing and able to provide written informed consent/assent for the trial.
7. Be at least 18 years of age on day of signing informed consent.
8. Have measurable disease based on RECIST 1.1.
9. Have provided tissue from an archival tissue sample or newly obtained core or excisional biopsy of a tumor lesion.
10. Have a performance status of 0 or 1 on the ECOG Performance Scale (See Appendix 12.3).
11. Demonstrate adequate organ function
12. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
13. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication (Reference Section 5.7.2). Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
14. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

1. Has disease which is amenable to radical treatment with surgery or radiation or a combination of treatments.
2. Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment.
3. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
4. Has had a prior monoclonal antibody within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
5. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
6. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
7. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment.
8. Has an active automimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjorgen's syndrome will not be excluded from the study.
9. Has evidence of interstitial lung disease
10. Has a history of non-infectious pneumonitis that required steroids, or has a history of active pneumonitis.
11. Has an active infection requiring systemic therapy.
12. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
13. Has known hypersensitivity to pembrolizumab (MK-3475) or its formulation.
14. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
15. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
16. Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
17. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
18. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
19. Has received a live vaccine within 30 days prior to the first dose of trial treatment.
20. Inability to swallow food or any condition of the upper gastrointestinal tract that precludes administration of oral medications.
21. Screening ECG with QTc interval > 480 milliseconds (corrected by Fridericia). In the event that a single QTc is >480 msec, the subject may enroll if the average QTc for 3 ECGs is < 480 msec.
22. Prior receipt of an IDO inhibitor.
23. Receipt of MAOIs within 21 days before first dose of study treatment.
24. History of serotonergic syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2021-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Giaccone, MD PhD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] He Y, Ramesh A, Gusev Y, Bhuvaneshwar K, Giaccone G. Molecular predictors of response to pembrolizumab in thymic carcinoma. Cell Rep Med. 2021 Sep 3;2(9):100392. doi: 10.1016/j.xcrm.2021.100392. eCollection 2021 Sep 21. PMID 34622229
- [Derived] Giaccone G, Kim C, Thompson J, McGuire C, Kallakury B, Chahine JJ, Manning M, Mogg R, Blumenschein WM, Tan MT, Subramaniam DS, Liu SV, Kaplan IM, McCutcheon JN. Pembrolizumab in patients with thymic carcinoma: a single-arm, single-centre, phase 2 study. Lancet Oncol. 2018 Mar;19(3):347-355. doi: 10.1016/S1470-2045(18)30062-7. Epub 2018 Jan 26. PMID 29395863

RESULTS

PARTICIPANT FLOW:
Groups:
- Pembrolizumab and Epacadostat: Pembrolizumab 200 mg intrvenoulsy every 3 weels
Period: Overall Study
Arm/Group | Pembrolizumab and Epacadostat
Started | 45
Completed | 40
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab and Epacadostat
Number analyzed (Participants) | 40
Age, Continuous [Median (Standard Deviation); unit: years] | 57 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 2
  White | 33
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: To measure response of all the participants to the drug at the end of the study.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Groups:
- Pembrolizumab: Pembrolizumab 200 mg intrvenoulsy every 3 weeks
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 40
Participants
  Complete Response | 1
  Partial response | 8
  Stable Disease | 21
  Progression | 10

2. Secondary Outcome: Progression-free Survival
Description: Time between start of treatment and tumor progression or death
Time Frame: 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 40
months | 4.2 [2.9 to 10.3]

3. Secondary Outcome: Overall Survival
Description: Time between start of treatment and death
Time Frame: 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 40
months | 24.9 [15.5 to NA] — Upper limit of the 95% confidence interval not reached

4. Secondary Outcome: Number of Participants With New-Onset Severe Adverse Events
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 40
Participants | 6

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Pembrolizumab and Epacadostat
All-Cause Mortality (participants affected / at risk) | 17/40
Serious Adverse Events (participants affected / at risk) | 6/40
Other Adverse Events (participants affected / at risk) | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab and Epacadostat (N=40)
Bullous pemphigoid (Immune system disorders) | 1
Polymoyositis (Musculoskeletal and connective tissue disorders) | 1
Hepatitis (Hepatobiliary disorders) | 1
Myocarditis (Cardiac disorders) | 2
Hyperglycemia (Endocrine disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab and Epacadostat (N=40)
Fatigue (General disorders) | 16
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
hypothyroidism (Endocrine disorders) | 5
hypokalemia (Metabolism and nutrition disorders) | 1
Elevated alkaline phosphatase (Metabolism and nutrition disorders) | 10
myocarditis (Cardiac disorders) | 2
AST elevation (Metabolism and nutrition disorders) | 16
Flu like (General disorders) | 2
ALT increased (Hepatobiliary disorders) | 10
Diarrhoea (Gastrointestinal disorders) | 9
Arthraglia (Musculoskeletal and connective tissue disorders) | 5
Fever (General disorders) | 5
Rhinitis (Immune system disorders) | 4
Anemia (Blood and lymphatic system disorders) | 4
Nausea (Gastrointestinal disorders) | 4
Rash (Immune system disorders) | 4
Myositis (Musculoskeletal and connective tissue disorders) | 3
Creatinine phosphokinase increased (Musculoskeletal and connective tissue disorders) | 3
Bilirubin increased (Hepatobiliary disorders) | 2
Blurred vision (Eye disorders) | 2
Dry mouth (Endocrine disorders) | 2
Hyperthyroidism (Endocrine disorders) | 2
Hyperurecemia (Endocrine disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 2
Amylase increased (Endocrine disorders) | 1
Dehydration (Endocrine disorders) | 1
Watering eyes (Endocrine disorders) | 1
Hyperglycemia (Endocrine disorders) | 1
Leucocytopenia (Blood and lymphatic system disorders) | 1
Lipased increased (Endocrine disorders) | 1
Facial swelling (Endocrine disorders) | 1
Palpitations (Cardiac disorders) | 1
skin disorders (Musculoskeletal and connective tissue disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-15): https://cdn.clinicaltrials.gov/large-docs/76/NCT02364076/Prot_SAP_000.pdf